CLINICAL TRIAL: NCT04349020
Title: Patient Reported Outcomes for Acute Asthma Care Treatment
Acronym: PROAACT
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Lin, Assistant Professor, Stanford University
Other Study IDs: GCO 17-2036; 1K23HL143042-01A1 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: Patient Reported Outcomes
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma affects 1 in every 12 persons in the U.S., resulting in 1.9 million ED visits annually; however, the impact of ED care on patient-reported outcomes after acute exacerbations is unknown. The proposed research will train a physician-scientist to develop a novel instrument to assess patient-reported outcomes after adult ED asthma visits, evaluate the association between ED clinical processes and patient-reported outcomes, and test the association between patient-reported outcomes and subsequent acute care utilization. The candidate will acquire skills in patient-centered research, instrument development and validation, and risk adjusted outcome measurement that will enable her transition to independence.

DETAILED DESCRIPTION:
This K23 award will enable the candidate, Michelle Lin, MD, MPH, MS, to become an independent physician scientist focused on developing, measuring and improving patient-reported outcomes for emergency department (ED) care of asthma and other acute cardiopulmonary conditions. Asthma affects 1 in every 12 persons in the U.S., resulting in 1.9 million ED visits annually; however, the impact of ED care on patient-reported outcomes after acute exacerbations is unknown-a gap which limits the evaluation of interventions to improve ED asthma care. Dr. Lin's proposed study aims to develop a patient-reported outcomes measure (PROM) for adult asthma patients seeking care in the ED, test the association between the quality of ED clinical care and patient-reported outcomes, and measure the association between patient-reported outcomes and subsequent acute care utilization. To achieve these goals, this proposal includes an integrated curriculum consisting of intensive mentorship and didactic coursework in patient-centered research, instrument development and validation including psychometric methods, geospatial techniques, outcome measurement, and risk adjustment. Her development and training activities also include building a research network of peers and collaborators, engaging with asthma patients in local communities, and participating in national scientific meetings. Dr. Lin has assembled a mentorship team of national leaders with expertise in patient-oriented asthma and emergency medicine research, patient engagement, instrument development, health care quality measurement, and outcome assessment. In her preliminary work, Dr. Lin has developed and pilot-tested candidate items for the novel Patient-Reported Outcomes for Acute Asthma Care and Treatment (PROAACT) instrument. During this K23, Dr. Lin will 1) evaluate the validity and reliability of the PROAACT instrument; 2) determine whether receiving more guideline-concordant ED care is associated with improved PROAACT responses; and 3) test the predictive validity of PROAACT responses with respect to subsequent ED visits and hospitalizations. Completion of this proposed project will result in a novel PROM for adult ED asthma patients and advance the understanding of how ED care impacts patient-reported outcomes, which will enable interventions to improve the quality of up to 1.9 million annual ED encounters for asthma. The proposed research and didactic plan will also facilitate Dr. Lin's transition to an independent clinical investigator focused on improving patient-reported outcomes for asthma and other cardiopulmonary conditions treated in ED settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English-speaking
* Prior diagnosis of asthma per the electronic health record
* Experiencing an ED visit for asthma as per ED clinician
* Medically appropriate for survey study as determined by treating ED clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients being discharged from ED after an acute exacerbation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcomes as measured by the PROAACT instrument | within 7-10 days of enrollment
  The study team will calculate patients' PROAACT scores and assess validity and reliability as a measure of quality after an ED visit asthma. the study team will compare PROAACT scores at the index visit (time of enrollment) and 7 days after enrollment. . Scale will be normalize on a Z-scale to produce a numeric value from 1-100 if validation is successful. A higher PROAACT score indicates improvement in patient-reported outcomes since the ED visit.

SECONDARY OUTCOMES:
Association between PROAACT scores and ED guideline adherence | within 7-10 days of enrollment
  The study team will assess ED clinician adherence to published guidelines for acute asthma care, and measure the association between guideline adherence and change in PROAACT scores. The study team hypothesizes patients receiving more guideline-concordant ED care will have greater improvement PROAACT scores at 7 days after the index ED visit.
Rate of acute care encounters | 30 days and 180 days after index ED visit (day of enrollment)
  (All-cause ED visit and/or hospitalization) Within 30 and 180 days after the index ED discharge. ED visits resulting in admission will count as one event.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lin, MD, MPH, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin MP, Vargas-Torres C, Schuur JD, Shi D, Wisnivesky J, Richardson LD. Trends and predictors of hospitalization after emergency department asthma visits among U.S. Adults, 2006-2014. J Asthma. 2020 Aug;57(8):811-819. doi: 10.1080/02770903.2019.1621889. Epub 2019 Jun 12. PMID 31112431
- [Derived] Lin MP, Gordon L, Richardson LD. Validating a Patient-Reported Outcome Measure to Improve Emergency Department Asthma Care: Protocol for an Observational Study. JMIR Res Protoc. 2025 May 29;14:e67195. doi: 10.2196/67195. PMID 40440691